CLINICAL TRIAL: NCT02021136
Title: Efficacy and Safety of Rebel Reliever Brace in Medial Femorotibial Knee Osteoarthritis. Phase 3, Multicenters, Randomised and Controlled Study With 2 Parallel Groups.
Brief Title: Efficacy and Safety of Rebel Reliever Brace in Patients With Symptomatic Medial Knee Osteoarthritis
Acronym: ROTOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A00613-42; 2013-A00613-42 (Other: ANSM number)
Record Dates: First submitted 2013-10-14; First posted 2013-12-27 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rebel reliever (Experimental): Rebel Reliever(R) knee brace + usual antalgic treatment + physical exercises recommendations.
  Interventions: Device: Rebel Reliever
- Control (Active Comparator): usual antalgic treatment + physical exercises recommendations.
  Interventions: Other: Control

INTERVENTIONS:
Device: Rebel Reliever — Rebel Reliever knee brace + usual antalgic treatment + physical exercises recommendations
  Arms: Rebel reliever
Other: Control — Usual antalgic treatment + physical exercises recommendations
  Arms: Control

SUMMARY:
The purpose of the study is to evaluate the superiority of Rebel Reliever® knee brace + standard treatment versus standard treatment alone in terms of last 24-hour pain relief after 6 weeks. in patients with medial knee osteoarthritis.

DETAILED DESCRIPTION:
The main criteria is the evaluation of global knee pain during the last 24 hours at D 49 after the inclusion.

The response to the treatment will be evaluated during the inclusion visit (V1/D0) and after 6 weeks of treatment, during the following visit (V3/D49).

The level of the global pain of the patient during the last 24 hours will be collected by investigators with a VAS (0 mm = no pain ; 100mm = maximun pain) at each visit.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female over 18 years
* BMI < or egal to 35kg/m2
* symptomatic gonarthrose defined by a recurrent pain to the walk on 30 days during the last 2 months before the inclusion with radiological findings (grade II to IV on Kellgren-Lawrence)
* diagnosis of medial femoro-tibial knee osteoarthrosis
* patient with global pain intensity during the last 24hours > or egal 40 mm (EVA) at the day of selection

Main Exclusion Criteria:

* femoro-patellar predominant arthrosis
* septic arthritis
* metabolic arthropathies
* chronical rheumatismal diseases
* other knee diseases
* symptomatic coxarthrosis
* controlateral gonathrosis with corticoids injections
* any other serious disease which may interfere with the results
* psychiatrics disorders
* skin lesions or dermal pathologies
* venous or arterial disorders
* sensitivity disorders in the lower limbs (diabetes mellitus..)
* paracetamol intolerance
* hyaluronic acid or corticosteroid intra-articular injection in the last month prior to inclusion
* on going knee viscosupplementation at inclusion
* slow acting OA drugs (if started in the last 2 months prior to inclusion)
* opioids, corticosteroids, or NSAIDs intake in the last 48 hours prior to inclusion
* pregnant women of with no contraception
* hepatic or renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Evolution of the last 24 hours knee pain (VAS) | Between Day 49 and Day 0

SECONDARY OUTCOMES:
Evolution of knee pain on movement (VAS) | Between Day 49 and Day 0
  Evaluation with Visual Analysis Scale
Evolution of Lequesne Algofunctional index score | Between D49 and Day 0
Responder rate according to OARSI-OMERACT criteria | At Day 49

OTHER OUTCOMES:
Percentage of patients with at least one adverse event or serious adverse event in each groups. | during the 6 weeks of brace wearing

CONTACTS AND LOCATIONS:
Overall Officials: Philippe THOUMIE, MD, Principal Investigator — Coordinator
Locations (1):
- Euraxi Pharma, Joué-lès-Tours, Bp 80325, France